CLINICAL TRIAL: NCT02569424
Title: Effect of PEEP and Trendelenburg on Ultrasound Size of Internal Jugular and Subclavian Veins: A Cross-over Randomized Controlled Study
Brief Title: Effect of PEEP and Trendelenburg on Ultrasound Size of Internal Jugular and Subclavian Veins
Acronym: PEEPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0246; 2015-A00606-43 (Registry Identifier: 2015-A00606-43)
Record Dates: First submitted 2015-09-24; First posted 2015-10-06 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Ventilated Patient in Intensive Care; Management of the Expiratory End-expiratory Pressure (PEEP) and Body Position
Keywords: PEEP level; Trendelenburg position; cross-sectional area of the jugular and subclavian veins; central venous catheter

ARMS (1):
- ventilated patients (Experimental): Patient's position (Supine or Trendelenburg strict -20°)
  Interventions: Behavioral: Patient's position

INTERVENTIONS:
Behavioral: Patient's position — Supine or Trendelenburg strict -20°)

SUMMARY:
There is no recommendation for the management of the positive end-expiratory pressure (PEEP) during setting of a central venous catheter (CVC) in a ventilated patient. Several non-randomized studies have investigated the cross-sectional area (AST) ultrasound minor axis for different pressure levels by evaluating a single vessel every time or by not displaying the right or left side in the evaluation. Another study showed that there could be unpredictable size differences between the 2 subclavian veins.

In ventilated patient, the PEEP, which is intrathoracic, will result in a decrease of venous return and thus possibly a superior vena cava dilation, located outside the pleura, depending on their capacitance. Different pressure levels showed an increase of AST with the increase of intra-thoracic pressure on certain veins, in a heterogeneous and not randomized manner.

The primary purpose of the study is to measure the effect of PEEP (0, 5, 10 or 15 cm H2O) and the patient's position (supine or Trendelenburg strict -15-20 °) on the cross-sectional area of the jugular and subclavian veins.

DETAILED DESCRIPTION:
There is no recommendation for the management of the positive end-expiratory pressure (PEEP) during setting of a central venous catheter (CVC) in a ventilated patient. Several non-randomized studies have investigated the cross-sectional area (AST) ultrasound minor axis for different pressure levels by evaluating a single vessel every time or by not displaying the right or left side in the evaluation. Another study showed that there could be unpredictable size differences between the 2 subclavian veins.

In ventilated patient, the PEEP, which is intrathoracic, will result in a decrease of venous return and thus possibly a superior vena cava dilation, located outside the pleura, depending on their capacitance. Different pressure levels showed an increase of AST with the increase of intra-thoracic pressure on certain veins, in a heterogeneous and not randomized manner.

The primary purpose of the study is to measure the effect of PEEP (0, 5, 10 or 15 cm H2O) and the patient's position (supine or Trendelenburg strict -15-20 °) on the cross-sectional area of the jugular and subclavian veins.

ELIGIBILITY:
Inclusion Criteria:

* Any patient ventilated in intensive care is eligible.
* Age ≥ 18 years
* Patient with stable hemodynamic status and Mean Blood Pressure (< 65 mmHg)
* Patient with registered social security number

Exclusion Criteria:

* clinical sign for a central venous thrombosis (unilateral edema ...).during echography screening before inclusion
* presence of a central line for more than 48 hours.
* Anechoic patient (checked during echography screening)
* History of cervical spine surgery.
* IntraCranial HyperTension
* patient in shock with hemodynamic instability and not stabilized
* patient treated by noradrenaline > 1 µg/kg/min
* patient or relative's refusal
* protected patients ≥ 18 years, minors, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The cross-sectional area of the jugular veins ( in cm2) | at baseline
  The cross-sectional area of the jugular veins ( in cm2) at the end of the intervention

SECONDARY OUTCOMES:
The cross-sectional area of the subclavian veins ( in cm2) | at baseline
  The cross-sectional area of the subclavian veins ( in cm2) at the end of the intervention
The antero-posterior diameter of the jugular veins (in mm) | at baseline
  The antero-posterior diameter of the jugular veins (in mm) at the end of the intervention
The antero-posterior diameter of the subclavian veins (in mm) | at baseline
  The antero-posterior diameter of the subclavian veins (in mm) at the end of the intervention
The distance between posterior and pleural lining of the jugular veins (in mm) | at baseline
  The distance between posterior and pleural lining of the jugular veins (in mm) at the end of the intervention
The distance between posterior and pleural lining of the subclavian veins (in mm) | at baseline
  The distance between posterior and pleural lining of the subclavian veins (in mm) at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France